CLINICAL TRIAL: NCT03939195
Title: OCTA Versus Structural OCT: Quantitative OCTA Biomarkers of Remission in Neovascular AMD
Brief Title: OCTA (Optical Coherence Angiography Tomography) Versus Structural OCT(Optical Coherence Tomography) in Neovascular AMD (Age Macular Degeneration)
Acronym: QUAOBARE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: QUAOBARE; 2018-A00948-47 (Other: ID-RCB)
Record Dates: First submitted 2019-01-11; First posted 2019-05-06 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Macular Degeneration Exudative Eye Left; Macular Degeneration Exudative Eye Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up — 4 follow-up visits with OCT Angiography and Structural OCT B

SUMMARY:
The objective is to find if there is a relationship between the Fractal Dimension, the gap, vascular density (VD), the surface, the span ratio and the status of the choroidal neovessels to adjust the interval between 2 intravitreal injections nor on the qualitative aspect of Optical Coherence Structural Tomography but also on quantified quantitative and objective values.

DETAILED DESCRIPTION:
This quantification is based on the analysis of fractal dimension (FD, without unit), lacunarity (Lac, without unit), vascular density (VD,%) and surface area of choroidal neovascular ( CNV, mm2).

The fractal dimension of a vascular structure corresponds to its degree of complexity. Fractals are models found in nature and biological systems that show self-similarity at different magnifications. It is obtained from the "box counting" method calculating the number of vascular segments contained in squares of varied size. Normal retinal vessels have a known and quantified complexity (FD = 1.7).

A neovascular tumor treated with anti-angiogenics will reduce vascular density, losing its random architecture; the investigators observe a return to a model standardized. NVCs have a random organization. The lower the FD, the more random the vascular architecture.

Lacunarity represents the texture or the homogeneity of a lesion, this one is heterogeneous when it is little vascularized and homogeneous if the vascularization is very dense. The lower the lake, the more homogeneous the lesion.

FD and Lac are obtained in Angiography Optical Coherence Tomography (OCTA) by the analysis of the hypersignal detected on the cut of the external retina.

The image is automatically binarised and skeletonized. NVC delineation is automatic and associated with automatic background noise processing. This software is fully automatic whose inter and intra grader reproducibility will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Man / woman over 50,
* Showing type 1 or type 2 CNV (choroidal neovessel) related to AMD during the second year of follow-up.
* Acceptance to participate in the protocol
* Affiliated to a social security scheme

Exclusion Criteria:

* Type III CNV related to AMD,
* Other cause of CNV
* Signal less than 80 decibel and detachment of pigment epithelium (PED) greater than 250 μm on structural OCT B.
* Protected Majors (Guardianship, Curator, Safeguard of Justice)
* Participation in another interventional research.
* Refusal to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to patients for whom intravitreal injections have already been performed for AMD-related choroidal neovascular vessels according to inclusion criteria over a period of four visits to TAE during the second year of therapeutic observation.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Fractal dimension (without unit) | 12 months
  Analysis of fractal dimension measured on OCT-A (Angiography Optical Coherence Tomography ) on 4 consecutive examinations.
Fractal lacunarity (without unit) | 12 months
  Analysis of lacunarity measured by OCT-A on 4 consecutive examinations.
Vascular density (%) | 12 months
  Analysis of vascular density measured by OCT-A on 4 consecutive examinations.
Vascular surface (micronm2) | 12 months
  Analysis of vascular surface measured by OCT-A on 4 consecutive examinations.

SECONDARY OUTCOMES:
Relationship between fractal dimension measured by OCT-A and choroidal neovascular (CNV) status | 12 months
  Investigation of a relationship between fractal dimension mesured on OCT-A and the status of choroidal neovessels
Relationship between fractal lacunarity measured by OCT-A and choroidal neovascular (CNV) status | 12 months
  Investigation of a relationship between fractal lacunarity and the status of choroidal neovessels
Relationship between vascular density measured by OCT-A and choroidal neovascular (CNV) status | 12 months
  Investigation of a relationship between vascula density and the status of choroidal neovessels
Relationship between vascular surface measured by OCT-A and choroidal neovascular (CNV) status | 12 months
  Investigation of a relationship between vascular surface and the status of choroidal neovessels

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHI Créteil, Créteil
  - Centre Bergouignan, Évreux
  - Centre d'exploration ophtalmologique de l'odéon, Paris

IPD SHARING:
Plan to Share IPD: No